CLINICAL TRIAL: NCT07134608
Title: Classical Popliteal Sciatic Block Versus Crosswise Approach for Popliteal Sciatic (CAPS) Block in Below Knee Surgery:A Randomised Control Trial
Brief Title: Comparing Classical Approach and Crosswise Approach to Popliteal Sciatic Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JEPUKM-JEP-2023-973
Record Dates: First submitted 2025-03-21; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-05

CONDITIONS: Popliteal Sciatic Nerve Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical Popliteal Sciatic Nerve Block (Active Comparator): Patients turned to the right or left lateral decubitus position, depending on which lower limb was planned for operation (i.e., right lateral decubitus if the operation was on the left lower limb and vice-versa). A pillow was placed between the lower limbs to facilitate block access and patient comfort. The classical popliteal sciatic block was done using a ultrasound machine with a high-frequency linear or low-frequency curvilinear probe placed 5-6 cm cranial to the popliteal fossa crease while identifying the bifurcation of the sciatic nerve. Skin infiltration with 5 ml of lignocaine 2% was performed using a 23G,followed by in-plane introduction of an 80 mm 22G block needle, aiming to penetrate the sciatic nerve sheath at the level of bifurcation, with placement confirmed using a nerve stimulator. After confirming negative aspiration for blood, 20 ml of Ropivacaine 0.5% was injected, and the spread of LA within the sheath was confirmed by ultrasound.
  Interventions: Procedure: Popliteal Plexus Block with 20 ml
- Crosswise Approach to Popliteal Sciatic Nerve (CAPS block) (Active Comparator): Patients in remained in the supine position. The CAPS block was performed using a similar Sonosite SII® ultrasound machine with a high-frequency linear or low-frequency curvilinear probe placed lateral to the thigh, 5-6 cm cranial to the popliteal fossa crease, while identifying the bifurcation of the sciatic nerve into the tibial and common peroneal nerves. Thereafter, the block proceeded similarly to patients in Group A, with 5 ml of lignocaine 2% for skin infiltration, in-plane introduction of the block needle aiming to penetrate the sciatic nerve sheath at the level of bifurcation and placement confirmed with a nerve stimulator, followed by injection of 20 ml of Ropivacaine 0.5% after confirming negative aspiration for blood. The spread of LA within the sheath was confirmed by ultrasound.
  Interventions: Procedure: Popliteal Plexus Block with 20 ml

INTERVENTIONS:
Procedure: Popliteal Plexus Block with 20 ml — Different position while blocking the popliteal sciatic nerve block

SUMMARY:
Sensory and motor innervation below the knee is provided mainly by the popliteal-sciatic nerve except for a variable area of the medial leg supplied by the saphenous nerve. Regional anaesthesia and analgesia for below knee surgery are frequently provided by blocking the popliteal sciatic nerve in the popliteal fossa. Popliteal sciatic block was first introduced around the 1970s and has emerged as a popular technique for below knee surgery despite other types of lower limb peripheral nerve block. This is contributed because popliteal fossa offers a superficial and accessible location for nerve blockade. This anatomical feature simplifies the procedure and may reduce the risk of complications such as vascular puncture or nerve injury.

Analgesia provided by the popliteal sciatic block lasts significantly longer than with ankle blocks. One of the reasons is administration of local anaesthetic agent at the popliteal fossa allows it to bathe the sciatic nerve before it bifurcates into the tibial and common peroneal nerves, leading to a more extensive and prolonged nerve blockade. Besides the sciatic nerve at the popliteal level is encased in a common epineural sheath, which can facilitate the spread of the anaesthetic and prolong its effect. The popliteal sciatic block can be performed as a single-shot technique or as a continuous infusion via a catheter The success rate of popliteal sciatic block is dependent on several variables, including the operator's skill, patient considerations, and surgical variables.

This study comparing between 2 approaches of popliteal sciatic nerve ie: classical approach and relatively new approach that is crosswise approach of popliteal sciatic nerve (CAPS) block.

ELIGIBILITY:
Inclusion Criteria:

* planned for either elective or non-elective unilateral below-knee surgery at HUKM
* patients aged 18 years and older and classified as physical status I, II, or III as dictated by the American Society of Anaesthesiologists (ASA)

Exclusion Criteria:

* included pregnant patients, those with a body mass index (BMI) ≥40 kg/m², contraindicated to peripheral nerve block (such as existing nerve injury to the limb intended for surgery), patient refusal, severe coagulopathy, local anaesthetic (LA) allergy, active infection at the intended block site, patients unable to provide a pain score using a verbal numerical rating scale (VNRS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Pain score during positioning and block performance | Time from positioning and block performance until completion of block (preoperative).
  Using verbal numerical rating scale (VNRS),ranging from 0 to 10, where 0 = no pain and 10 = the worst pain imaginable.

SECONDARY OUTCOMES:
Fentanyl consumption | On operative day until post operative day 1
  Aliquots of intravenous (IV) fentanyl (25-50 micrograms) were given if the patient experienced pain with a VNRS ≥4 during positioning or block performance.
Onset of block | Immediately after block completion until 30 minutes after.
  Adequacy of the block was assessed at 5-minute intervals based on the loss of pain sensation to pin prick with a 23G (B. Braun®) needle in the distribution of the popliteal sciatic nerve (measure in minutes).
Failure rate | 30 minutes after block completion
  Persistent pain sensation after 30 minutes over popliteal sciatic nerve distribution
Patient's satisfaction | One day after procedure.
  Patient satisfaction with the block was assessed using a five-point Likert scale (1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied, 5 = very satisfied).
Complications | On operative day until post operative day 1
  Such as hematoma, L.A toxicity, or persistent numbness/weakness lasting more than 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Canselor Tuanku Muhriz, Kuala Lumpur, Kuala Lumpur, Malaysia